CLINICAL TRIAL: NCT03017209
Title: Study on a Locally Prepared Food Supplement to Support Growth and Brain Health
Brief Title: Locally Prepared Supplement to Support Growth and Brain Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Massachusetts General Hospital (Other); Global Food & Nutrition Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12356
Record Dates: First submitted 2016-12-17; First posted 2017-01-11 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Malnutrition, Child; Cognitive Function
MeSH Terms: conditions — Child Nutrition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Locally-prepared bar (Experimental): The bar is similar to one tested recently in a pilot study and is a locally prepared bar designed to facilitate growth and cognitive development. It will provide 300 kcal/day and will have ≈20-30% of energy from protein (of which 25-50% is from an animal protein source), 20-35% from total carbohydrate and ≈40-60% from fat. The bar will be fortified with vitamins and minerals to meet USAID recommendations for moderate malnutrition and Dietary Reference Intake recommendations for at-risk and healthy children of the ages studied, and at the same time will not exceed Upper Level nutrient recommendations for any micronutrient. Ingredients in the bar will be a combination of local products and imported shelf-stable ingredients.
  Interventions: Dietary Supplement: Locally-prepared bar
- USAID Corn Soy Blend Plus (Active Comparator): The usual-intervention condition will be 300 kcal/day of USAID Corn Soy Blend Plus cooked in the usual manner with fortified vegetable oil (10:3 ratio) and sugar. The community health workers or other designated villagers will prepare the supplement freshly each intervention day using locally accepted standards for hygiene, and a quality control process for ratios of ingredients assigned by the research team to ensure consistent composition.
  Interventions: Dietary Supplement: USAID Corn Soy Blend Plus
- Locally-purchased rice (Placebo Comparator): The placebo condition will be 300 kcal/day of locally-purchased rice cooked with a small amount of oil (10:2 ratio), which mimics the usual breakfast of children in this region. The community health workers or other designated villagers will prepare the rice freshly each intervention day using locally accepted standards for hygiene, and a quality control process for ratios of ingredients assigned by the research team to ensure consistent composition.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Locally-prepared bar — School children in first grade will receive their supplement 5 days a week in the morning before school starts. Younger children will receive the supplement 5 days a week in the morning at the community health center, distributed by community health workers. The teachers and community health workers will record amount of supplement consumption daily during the study, and will report the information weekly to the local research team throughout the intervention period.
  Arms: Locally-prepared bar
Dietary Supplement: USAID Corn Soy Blend Plus — School children in first grade will receive their supplement 5 days a week in the morning before school starts. Younger children will receive the supplement 5 days a week in the morning at the community health center, distributed by community health workers. The teachers and community health workers will record amount of supplement consumption daily during the study, and will report the information weekly to the local research team throughout the intervention period.
  Arms: USAID Corn Soy Blend Plus
Other: Placebo — School children in first grade will receive their supplement 5 days a week in the morning before school starts. Younger children will receive the supplement 5 days a week in the morning at the community health center, distributed by community health workers. The teachers and community health workers will record amount of supplement consumption daily during the study, and will report the information weekly to the local research team throughout the intervention period.
  Other Names: Locally-purchased rice
  Arms: Locally-purchased rice

SUMMARY:
This study is a randomized controlled trial with a main goal to assess the effects of a locally-prepared food for prevention of malnutrition and stunting, in comparison with standard village practices and also a widely available aid food supplement in 8-12 villages in Guinea-Bissau. The supplement intervention will be for 24-30 weeks. The primary outcome will be cognitive tests of executive function. Secondary outcomes will be changes in standard anthropometric benchmarks of growth, hemoglobin and skin carotenoids in young children living in villages in rural Guinea-Bissau. This is a within-village randomization at the level of the family, and all children will receive a dietary intervention.

DETAILED DESCRIPTION:
Up to 1050 children aged 15 months to 6.99 years, and older children if in 1st grade elementary school, in 8-12 villages in the Oio and Cachau regions of Guinea-Bissau will be recruited for this study along with their maternal caregiver and father. Child ages will be based on the official birth records which families possess. The mothers/primary caregivers and fathers of the children will also be recruited for simple outcome assessments. Villages will be a convenience sample chosen from villages within the network of our local research partner International Partnership for Human Development. Each village in this region has one school and one community health center per village, which will be involved in supplement distribution and some outcome assessments.

Families with enrolling children will be randomized within 8-12 villages to receive 1 of 3 supplements and if any family (defined based on the father of the children since this is a polygamous community) has more than one enrolling child all those children will be randomized to the same supplement arm.

* One supplement will be the locally-prepared bar
* One will be an isocaloric amount of porridge prepared with USAIDs Corn Soy Blend Plus, prepared as recommended in a 10:3 ratio with fortified vegetable oil.
* One supplement will be an isocaloric amount of cooked rice with vegetable oil, which is the typical local breakfast.

Villagers will be informed of the randomization after baseline testing is complete.

Following baseline measurements in children of anthropometry and body composition, grip strength, cognition, hemoglobin, and skin carotenoids, children will receive their intervention for 24-30 weeks and the same measurements taken at baseline will be repeated during the last study week. The flexible end data is given to accommodate the local rainy season and its impact on transportation. Please note that cell phone access to villages is not influenced by local weather, thus communication regarding safety issues with community health workers will remain possible throughout the entire trial.

Addendum: The pre-planned primary method of analysis was a per-protocol analysis, predefined as children consuming ≥75% of their supplement. However, a clerical error in this clinical trial registration did not describe this predetermined focus on a per-protocol population. The registration implies an intention-to-treat (ITT) analysis by default. Investigators therefore revised our analytical approach to designate the ITT cohort as the primary cohort of interest. The secondary cohort of interest is the predefined per-protocol cohort (children consuming ≥75% of their supplement).

ELIGIBILITY:
Inclusion Criteria:

* Parent or legal guardian provides consent for all children <7 years and the parent plus the child provide consent for any child > 7 years.
* Age 15 months to 6.99 years old or any age enrolled in first grade in the same village.
* The family plans to remain in the village for the duration of the study (up to 30 weeks) based on self-report by a parent;
* The child does not have any known food allergies as reported by the mother or guardian.

Exclusion Criteria: If any child is identified as malnourished at baseline, defined as a mid-upper arm circumference in the red zone of the paper tape, the child will be excluded from the study due to malnutrition, and the parents will be advised to take the child to the nearest malnutrition clinic.

Ages: 15 Months to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1059 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change in cognitive function measured using executive functions tasks in children ages 15 months to 3 years | baseline and 24-30 weeks after baseline testing

SECONDARY OUTCOMES:
Hemoglobin | baseline and 24-30 weeks after baseline testing
Changes in z-scores for weight (WAZ) | baseline and 24-30 weeks after baseline testing
Changes in z-scores for height (HAZ) | baseline and 24-30 weeks after baseline testing
Cognitive tests for children >3 years old | baseline and 24-30 weeks after baseline testing
  Looking to see changes in executive function who attend supplement distribution at least 75% of the days it is offered.
Mid-upper arm circumference | baseline and 24-30 weeks after baseline testing
Cerebral blood flow | baseline and 24-30 weeks after baseline testing
  By infrared spectroscopy
% Lean tissue and lean growth | baseline and 24-30 weeks after baseline testing
Changes in weight for height Z scores | baseline and 24-30 weeks after baseline testing

OTHER OUTCOMES:
Carotenoids | baseline and 24-30 weeks after baseline testing
  By Resonance Raman Spectroscopy
Grip strength | baseline and 24-30 weeks after baseline testing
  Using a dynamometer
Weight of female-caregivers and fathers | baseline and 24-30 weeks after baseline testing
Head circumference of child | baseline and 24-30 weeks after baseline testing
Height of female-caregivers and fathers | baseline and 24-30 weeks after baseline testing
Mid upper arm circumference of female caregivers | baseline and 24-30 weeks after baseline testing

CONTACTS AND LOCATIONS:
Overall Officials: Susan B Roberts, PHD, Principal Investigator — Tufts University
Locations (1):
- International Partnership for Health Development, Bissau, Guinea-Bissau

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roberts SB, Franceschini MA, Silver RE, Taylor SF, de Sa AB, Co R, Sonco A, Krauss A, Taetzsch A, Webb P, Das SK, Chen CY, Rogers BL, Saltzman E, Lin PY, Schlossman N, Pruzensky W, Bale C, Chui KKH, Muentener P. Effects of food supplementation on cognitive function, cerebral blood flow, and nutritional status in young children at risk of undernutrition: randomized controlled trial. BMJ. 2020 Jul 22;370:m2397. doi: 10.1136/bmj.m2397. PMID 32699176
- [Derived] Roberts SB, Franceschini MA, Krauss A, Lin PY, de Sa AB, Co R, Taylor S, Brown C, Chen O, Johnson EJ, Pruzensky W, Schlossman N, Bale C, Wu KT, Hagan K, Saltzman E, Muentener P. A Pilot Randomized Controlled Trial of a New Supplementary Food Designed to Enhance Cognitive Performance during Prevention and Treatment of Malnutrition in Childhood. Curr Dev Nutr. 2017 Nov;1(11):e000885. doi: 10.3945/cdn.117.000885. Epub 2017 Oct 12. PMID 29658962